CLINICAL TRIAL: NCT01639131
Title: A Multi-institutional Open Label, Trial Evaluating the Efficacy of Gemcitabine and Docetaxel in Patients With Relapsed or Refractory Metastatic Colorectal Adenocarcinoma With Methylated CHFR and/or Microsatellite Instability Phenotype
Brief Title: Gemcitabine and Docetaxel in Patients With Relapsed or Refractory Metastatic Colorectal Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1214; NA_00069666 (Other: JHMIRB)
Record Dates: First submitted 2012-07-09; First posted 2012-07-12 (Estimated); Results first posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Colorectal Adenocarcinoma
Keywords: Gemcitabine; Docetaxel; Filgrastim; Pegfilgrastim; Colorectal Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; Docetaxel; Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine and Docetaxel (Experimental): Patients were treated with gemcitabine 800 mg/m2 on days 1 and 8 and docetaxel 70 mg/m2 on day 8 of each 21-day cycle. Patients received filgrastim (granulocyte colony-stimulating factor [G-CSF]) on days 9 through 15 or pegfilgrastim 6 mg on day 9 or 10 of each cycle. Patients were treated until disease progression or unacceptable adverse events (AEs), or withdrawn of the consent.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Drug: Filgrastim or Pegfilgrastim

INTERVENTIONS:
Drug: Gemcitabine — intravenous gemcitabine 800mg/m2 on days 1 and 8
Drug: Docetaxel — intravenous docetaxel 70mg/m2 on day 8 of each 21 day cycle
Drug: Filgrastim or Pegfilgrastim — filgrastim (granulocyte colony-stimulating factor [G-CSF]) on days 9 through 15 or pegfilgrastim 6 mg on day 9 or 10 of each cycle

SUMMARY:
The primary goal of the trail was to determine the efficacy of combining Gemcitabine and Docetaxel in treatment of metastatic colorectal cancer with CHFR and/or Microsatellite Instability (MSI) phenotype.

DETAILED DESCRIPTION:
This was an open-label, multicenter, trial. Enrolled patients received an intravenous combination of gemcitabine 800 mg/m2 on days 1 and 8 and docetaxel 70 mg/m2 on day 8 of each 21-day cycle. Patients received filgrastim (granulocyte colony-stimulating factor [G-CSF]) on days 9 through 15 or pegfilgrastim 6 mg on day 9 or 10 of each cycle. Patients were treated until disease progression or unacceptable adverse events (AEs), or withdrawn of the consent.

Patients underwent safety evaluations and monitoring for adverse events for each cycle.

Disease assessments (computed tomography or magnetic resonance imaging) were performed at baseline and then every 6 weeks. Response was evaluated according to the RECIST version1.1.

Patients who discontinue treatment will be monitored for overall survival.

ELIGIBILITY:
Inclusion:

* Patients must have histologically or cytologically confirmed metastatic or unresectable adenocarcinoma of the colon or rectum.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Patients must be either intolerant or refractory to one or more standard line(s) of chemotherapy treatment prior to enrollment. Toxicity from prior regimens must be resolved to less than or equal to grade 1 prior to enrollment. Patients with grade 2 neurotoxicity may be enrolled on a case by case basis at the discretion of the principle investigator. Patients should be off all treatment for at least 4 weeks prior to trial enrollment.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of gemcitabine in combination with docetaxel in patients <18 years of age with colorectal adenocarcinoma, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status 0 or 1 (Karnofsky >70%, see Appendix A).
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function.

Additional eligibility criteria:

* Microsatellite instability phenotype of archival tissue biopsy determined by treating institution by PCR and IHC assay
* Methylation CHFR gene promoter in archival tissue biopsy
* As gemcitabine and docetaxel are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine or docetaxel.
* Patients receiving any medications or substances that are inhibitors or inducers of CYP 3A4 are ineligible. Lists including medications and substances known or with the potential to interact with the cytochrome 450 3A4 isoenzyme are provided in appendix C.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects of study medications. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with gemcitabine and docetaxel breastfeeding should be discontinued if the mother is treated. These potential risks may also apply to other agents used in this study including supportive medications.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with gemcitabine and docetaxel. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-09-10 (Actual); Primary Completion 2016-10-03 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer Azad, Principal Investigator — SKCCC at JHMI
Locations (3):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Center for Cancer Research, NCI, Bethesda, Maryland
- VU Medisch Centrum, Amsterdam, Netherlands

REFERENCES:
- [Derived] Baretti M, Karunasena E, Zahurak M, Walker R, Zhao Y, Pisanic TR 2nd, Wang TH, Greten TF, Duffy AG, Gootjes E, Meijer G, Verheul HMW, Ahuja N, Herman JG, Azad NS. A phase 2 trial of gemcitabine and docetaxel in patients with metastatic colorectal adenocarcinoma with methylated checkpoint with forkhead and ring finger domain promoter and/or microsatellite instability phenotype. Clin Transl Sci. 2021 May;14(3):954-963. doi: 10.1111/cts.12960. Epub 2021 Apr 3. PMID 33811727
- See also: A phase 2 trial of gemcitabine and docetaxel in patients with metastatic colorectal adenocarcinoma with methylated checkpoint with forkhead and ring finger domain promoter and/or microsatellite instability phenotype Marina Baretti 1, Enusha Karunasena 1, — https://pubmed.ncbi.nlm.nih.gov/33811727/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine and Docetaxel: Patients received intravenous gemcitabine 800mg/m2 on days 1 and 8 and docetaxel 70mg/m2 on day 8 of each 21 day cycle. Patients received filgrastim (G-CSF) on days 9 through 15 or pegfilgrastim 6mg on day 9 or 10 of each cycle.
  Gemcitabine: intravenous gemcitabine 800mg/m2 on days 1 and 8
  Docetaxel: docetaxel 70mg/m2 on day 8 of each 21 day cycle
  Filgrastim or Pegfilgrastim: filgrastim (G-CSF) on days 9 through 15 or pegfilgrastim 6mg on day 9 or 10 of each cycle
Period: Overall Study
Arm/Group | Gemcitabine and Docetaxel
Started | 6
Completed | 0
Not Completed | 6
Not completed — Disease Progression | 6

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Docetaxel
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: The Response Rate is defined as the number of patients achieving a complete response (CR) or partial response (PR) based on the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). CR = disappearance of all target lesions, PR is =>30% decrease in sum of diameters of target lesions, progressive disease (PD) is >20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: 9 months
Measure: Number; unit: participants
Arm/Group | Gemcitabine and Docetaxel
Number analyzed (Participants) | 6
participants | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. PFS is defined as the number of months from the date of first dose of study drug to disease progression (progressive disease [PD] or relapse from complete response [CR] as assessed using RECIST 1.1 criteria) or death due to any cause. Per RECIST 1.1 criteria, CR = disappearance of all target lesions, Partial Response (PR) is =>30% decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20% increase in sum of diameters of target lesions, Stable Disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Time Frame: 9 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine and Docetaxel
Number analyzed (Participants) | 6
months | 1.79 [1.28 to NA] — The upper limit of the KM curve has not reached 50%, therefore there is no estimate for the upper confidence limit on the median

3. Secondary Outcome: Overall Survival With Gemcitabine and Docetaxel Combination Therapy
Description: Overall survival is the time from the start of first dose of study drug to death. OS will be measured from date of first dose of a study drug until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: 62 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine and Docetaxel
Number analyzed (Participants) | 6
months | 15.67 [4.24 to NA] — The upper limit of the KM curve has not reached 50%, therefore there is no estimate for the upper confidence limit on the median

ADVERSE EVENTS:
Time Frame: Survival was monitored for up to 62 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored for 9 months.
Description: During the survival follow-up portion of the trial, participants were evaluated for all-cause mortality past the time frame of treatment and the assessment of Serious and Other (Not Including Serious) Adverse Events.
Arm/Group | Gemcitabine and Docetaxel
All-Cause Mortality (participants affected / at risk) | 4/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Docetaxel (N=6)
fever (Investigations) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
neuropathic fever (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine and Docetaxel (N=6)
Lymphocyte count decreased (Investigations) | 3 (14)
Anemia (Blood and lymphatic system disorders) | 3 (12)
White blood cell decreased (Investigations) | 3 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (6)
Neutrophil count decreased (Investigations) | 1 (5)
Platelet count decreased (Investigations) | 4 (5)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (5)
Alkaline Phosphatase increased (Investigations) | 1 (1)
Alanine Aminotransferase increased (Investigations) | 1 (1)
Fever (General disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)
Thrombus (Vascular disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Diarhhea (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (4)
Edema Face (General disorders) | 1 (2)
Edema limbs (General disorders) | 2 (2)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Localized Edema (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (5)
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT01639131/Prot_SAP_000.pdf